CLINICAL TRIAL: NCT06046339
Title: Evolution of Left Ventricular Ejection Fraction After Treatment of Out-of-hospital Cardiac Arrest by Extracorporeal Cardiopulmonary Resuscitation
Brief Title: Left Ventricular Ejection Fraction in Cardiac Arrest Survivors Treated With Extracorporeal Cardiopulmonary Resuscitation
Acronym: FEVGECMO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230308
Record Dates: First submitted 2023-09-04; First posted 2023-09-21 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Out-of-Hospital Cardiac Arrest; Extracorporeal Cardiopulmonary Resuscitation
Keywords: Out-of-Hospital Cardiac Arrest; Extracorporeal cardiopulmonary resuscitation; Left ventricular function; Left ventricular ejection fraction
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients hospitalized at Necker Hospital for an extra-hospital cardiac arrest between January 1, 2015 and October 31, 2019.
  Interventions: Other: Collection of data from the patient's medical file

INTERVENTIONS:
Other: Collection of data from the patient's medical file — Collection of data from the patient's medical file.

SUMMARY:
Extra-hospital cardiac arrest is a major public health problem, with approximately 46,000 cases per year. Nearly 71% of the patients for whom resuscitation was initiated did not present a return of spontaneous circulation on scene and only 29% were transported alive to the hospital. In this context, extracorporeal cardiopulmonary resuscitation (ECPR) by veno-arterial extracorporeal membrane oxygenation has been developed as a second line of treatment according to the latest international guidelines. The selection of eligible patients as well as the timing of initiation of ECPR has long been controversial, but expert recommendations have recently been published.

After an out-of-hospital cardiac arrest of cardiological cause, an early ventricular dysfunction has been previously described, more particularly in hemodynamically unstable patients. This dysfunction was associated with greater early in-hospital mortality. There are few data on the medium-term course of left ventricular dysfunction and the largest study addressing this question showed that the severity of left ventricular involvement was associated with greater long-term morbidity and mortality. However, it also found that left ventricular ejection fraction was partially reversible in 29% of the study population.

It seems so far, the medium-term evolution of left heart dysfunction had not been described in the context of refractory extra-hospital cardiac arrest treated by ECPR. However, these patients are particularly severe, hemodynamically unstable and potentially at risk of developing long-term sequelae.

DETAILED DESCRIPTION:
Extra-hospital cardiac arrest is a major public health problem, with approximately 46,000 cases per year. Nearly 71% of the patients for whom resuscitation was initiated did not present a return of spontaneous circulation on scene and only 29% were transported alive to the hospital. In this context, extracorporeal cardiopulmonary resuscitation (ECPR) by veno-arterial extracorporeal membrane oxygenation has been developed as a second line of treatment according to the latest international guidelines. The selection of eligible patients as well as the timing of initiation of ECPR has long been controversial, but expert recommendations have recently been published.

After an out-of-hospital cardiac arrest of cardiological cause, an early ventricular dysfunction has been previously described, more particularly in hemodynamically unstable patients. This dysfunction was associated with greater early in-hospital mortality. There are few data on the medium-term course of left ventricular dysfunction and the largest study addressing this question showed that the severity of left ventricular involvement was associated with greater long-term morbidity and mortality. However, it also found that left ventricular ejection fraction was partially reversible in 29% of the study population.

It seems so far, the medium-term evolution of left heart dysfunction had not been described in the context of refractory extra-hospital cardiac arrest treated by ECPR. However, these patients are particularly severe, hemodynamically unstable and potentially at risk of developing long-term sequelae.

The research focuses on the evolution of left ventricular function at 28 and 90 days after an out-of-hospital refractory cardiac arrest treated with ECPR as well as describing the survival rate at 28 and 90 days for these patients.

The expected results are to demonstrate that the left ventricular function, described through the left ventricular ejection fraction, is seriously affected in the population studied without signs of reversibility. These patients would therefore need close cardiological follow-up and to be integrated into a dedicated care pathway.

ELIGIBILITY:
Inclusion Criteria:

* Implementation of an extracorporeal membrane oxygenation (ECMO) following an acute coronary syndrome (ACS) defined for the purposes of the study by the existence of at least one of the following criteria: ST segment elevation or depression on the electrocardiogram associated with chest pain and elevated plasma troponin levels; a coronary angiography showing at least one significant coronary lesion and/or having required revascularization. Confirmation of an ischemic etiology by post-mortem examination. A coronary lesion is considered significant if it is described by the cardiologist as: acute and responsible for a reduction in the caliber of the artery strictly greater than 70% and less than 99% for a severe stenosis, and 100% for a complete stenosis.
* Patients hospitalized at Necker Hospital for pre-hospital cardiac arrest between January 1, 2015 and October 31, 2019.
* Sending to living patients of the study information note, a period of one month is given to the patients to oppose the use of their data for the study.

Exclusion Criteria:

* Extracorporeal membrane oxygenation implementation outside the context of refractory out-of-hospital cardiac arrest
* In-hospital cardiac arrests
* Obvious non-cardiological cause of cardiac arrest
* Cardiac arrests unrelated to acute coronary syndrome
* Cardiac arrests for which no etiology has been found
* Patients opposed to the use of their data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized at Necker Hospital for an extra-hospital cardiac arrest between January 1, 2015 and October 31, 2019.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-05-04 (Actual); Study Completion 2024-05-04 (Actual)

PRIMARY OUTCOMES:
Quantitative Assessment of Left Ventricular Ejection Fraction Using Ultrasound Values, 28 Days After Cardiac Arrest | At 28 days after cardiac arrest
  Left ventricular ejection fraction value at 28 days after out-of-hospital cardiac arrest treated by extracorporeal cardiopulmonary resuscitation.

SECONDARY OUTCOMES:
Quantitative Assessment of Left Ventricular Ejection Fraction Using Ultrasound Values, 90 Days After Cardiac Arrest | At 90 days after cardiac arrest
  Left ventricular ejection fraction value at 90 days after out-of-hospital cardiac arrest treated by extracorporeal cardiopulmonary resuscitation.
Survival | At 28 and at 90 days after cardiac arrest
  Survival rate at 28 days and at 90 days after out-of-hospital cardiac arrest treated by extracorporeal cardiopulmonary resuscitation.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Herlé RAPHALEN, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khoury J, Soumagnac T, Vimpere D, El Morabity A, Hutin A, Raphalen JH, Lamhaut L. Long-term heart function in refractory out-of-hospital cardiac arrest treated with prehospital extracorporeal cardiopulmonary resuscitation. Resuscitation. 2025 Feb;207:110449. doi: 10.1016/j.resuscitation.2024.110449. Epub 2024 Nov 30. PMID 39622448
- [Background] Luc G, Baert V, Escutnaire J, Genin M, Vilhelm C, Di Pompeo C, Khoury CE, Segal N, Wiel E, Adnet F, Tazarourte K, Gueugniaud PY, Hubert H; On behalf GR-ReAC. Epidemiology of out-of-hospital cardiac arrest: A French national incidence and mid-term survival rate study. Anaesth Crit Care Pain Med. 2019 Apr;38(2):131-135. doi: 10.1016/j.accpm.2018.04.006. Epub 2018 Apr 21. PMID 29684654
- [Background] Registre électronique des arrêts cardiaques. Données du 1 er juillet 2011 au 31 mai 2021. Adresse : https://registreac.org/.
- [Background] Soar J, Bottiger BW, Carli P, Couper K, Deakin CD, Djarv T, Lott C, Olasveengen T, Paal P, Pellis T, Perkins GD, Sandroni C, Nolan JP. European Resuscitation Council Guidelines 2021: Adult advanced life support. Resuscitation. 2021 Apr;161:115-151. doi: 10.1016/j.resuscitation.2021.02.010. Epub 2021 Mar 24. PMID 33773825
- [Background] Hutin A, Abu-Habsa M, Burns B, Bernard S, Bellezzo J, Shinar Z, Torres EC, Gueugniaud PY, Carli P, Lamhaut L. Early ECPR for out-of-hospital cardiac arrest: Best practice in 2018. Resuscitation. 2018 Sep;130:44-48. doi: 10.1016/j.resuscitation.2018.05.004. Epub 2018 May 5. PMID 29738799
- [Background] Gupta A, Gupta A, Saba S. Change in myocardial function after resuscitated sudden cardiac arrest and its impact on long-term mortality and defibrillator implantation. Indian Pacing Electrophysiol J. 2019 Jul-Aug;19(4):150-154. doi: 10.1016/j.ipej.2019.04.005. Epub 2019 Apr 22. PMID 31022454